CLINICAL TRIAL: NCT03941158
Title: Cohabitation Patterns and Incidence of Known and Suspected Sexually Transmitted Diseases
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Principal Investigator, Christian Erikstrup, Professor, Chief Physician, Aarhus University Hospital
Other Study IDs: 2015-57-0102
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Cohabitation Patterns; Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of infectious agents associated with risks of malignant hematologic diseases is non-negligible and include both viruses and bacteria.

The various organisms affect cancer risk either directly by transforming susceptible cells, through chronic antigenic stimulation or by hampering immune function in other ways conducive of cancer development.

Suspicion of an infectious cancer origin may arise because of clustering with other conditions (e.g. immune deficiency), specific environments or settings (e.g. geographic locales) or with exposures (e.g. blood transfusions).

In this context, relatively few studies have addressed clustering of diseases among spouses to generate hypotheses about the relative contributions of environmental and genetic factors to the risk of individual cancer types.

As a prelude to such an exercise aiming specifically at malignant hematologic diseases, we will test an algorithm characterising cohabitation patterns in the Danish population to assess the risk of sexually transmitted diseases in analyses of register data.

Such information will also be relevant to current guidelines for blood donor deferral policies. Specifically, because of the so-called precautionary principle all blood donations are extensively tested for infectious agents and transfusion of blood now carries an extremely low risk of transmission of HIV, hepatitis B and C. The residual risk of HIV transmission in Denmark is estimated to 1:10,000,000 transfusions. However, several deferral criteria have existed for years without studies to prove their relevance.

Aim: To compare the incidence of both known and suspected sexually transmitted diseases between different cohabitation patterns in the Danish population.

Perspectives: The study results can be used to leverage changes in deferral rules in the Danish blood banks to accommodate strong wishes from stakeholders to avoid the perceived discrimination of various minorities. The study can thus have important ethical and political consequences.

ELIGIBILITY:
Inclusion Criteria:

* All citizens in Denmark

Exclusion Criteria:

* Institutionalized individuals

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In Denmark, every citizen is registered with a unique identification number in the Civil Registration System. Adult persons (18 years or older) who resided in Denmark for any period between 1 April 1968 and primo 2018 will be identified and linked to national health registers by using the unique identification number.
  Different living arrangements can be defined by using an address-based algorithm to identify each citizen's complete day-by-day cohabitation or marital status history.
Sampling Method: Probability Sample
Enrollment: 5000000 (Actual)
Dates: Start 1968-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Sexually transmitted diseases | 1977 - 2018
  The diseases will be identified by using the Danish National Patient Register (NPR). Diagnostic information is based on the International Classification of Diseases, Eight and Tenth Revision (ICD-8 and ICD-10).
HIV, syphilis, and gonorrhea | 2005 - 2018
  HIV, syphilis, and gonorrhea will be identified by registration in the Mandatory disease notification system administrated by Statens Serums Institut (SSI), Denmark.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Erikstrup, Professor, Chief Physician, Principal Investigator — Aarhus University Hospital